CLINICAL TRIAL: NCT03997370
Title: Assessment of Carboplatin Clearance Predictors: A PK Study on NCI-Sponsored Clinical Trials or Standard of Care Treatments Using Carboplatin
Brief Title: Evaluation of Dosing Procedures of Chemotherapy Treatment (Carboplatin) With the Contrast Agent Iohexol
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GY022; NCI-2019-04008 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY022 (Other: NRG Oncology); NRG-GY022 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2019-06-24; First posted 2019-06-25 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Malignant Solid Neoplasm
MeSH Terms: interventions — Specimen Handling; Carboplatin; Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (iohexol, standard care carboplatin, blood samples) (Experimental): Patients receive iohexol IV over 30-60 seconds. Patients then receive standard of care carboplatin IV. Patients also undergo collection of 7-8 blood samples for analysis.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Iohexol

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Iohexol — Given IV
  Other Names: Omnipaque

SUMMARY:
This trial studies how well iohexol works in helping doctors calculate the dose of carboplatin given to patients with cancer. Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Understanding how to best calculate the dose of carboplatin given to patients with cancer may help doctors learn how to improve the use of carboplatin in the future.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the success of targeting a carboplatin area under the curve (AUC) with our current approach to dosing carboplatin.

II. Assess the performance of Cockcroft-Gault (CG), four-variable Modification of Diet in Renal Disease (MDRD-4), and Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) based on isotope dilution mass spectrometry (IDMS) calibrated serum creatinine in predicting measured glomerular filtration rate (mGFR) in patients with cancer.

III. Define the relationship of mGFR and carboplatin clearance in patients with cancer.

SECONDARY OBJECTIVES:

I. Evaluate the divergence of estimated (e)GFR from mGFR based on patient demographic and other characteristics, thus identifying those most likely to benefit from determination of mGFR over use of eGFR.

II. Determine the success rate of achieving the target carboplatin AUC in patients in whom the carboplatin dose is capped.

III. Evaluate the relationship between carboplatin exposure and toxicity. IV. Assess the ability of markers other than creatinine in pre-treatment serum to better estimate kidney function in patients with cancer.

OUTLINE:

Patients receive iohexol intravenously (IV) over 30-60 seconds. Patients then receive standard of care carboplatin IV. Patients also undergo collection of 7-8 blood samples for analysis.

After completion of study, patients are followed up for 3-4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the psychological ability and general health that permits completion of the study requirements and required follow up
* For men who are sexually active, the need for use of medically acceptable contraception will be dictated by the primary treatment plan/protocol

  * Study accrual was closed to women on 08/18/2021 and accrual is now only open to males in order to meet accrual goals and study objectives. (11-AUG-2021)
* Male sex
* Any patients who will receive treatment with intravenous carboplatin (any AUC, any cycle) on a National Cancer Institute (NCI)-sponsored National Clinical Trial Network (NCTN)-, Experimental Therapeutics Clinical Trials Network (ETCTN)-, trial, local trial, or through standard of care
* Age >= 18
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry

Exclusion Criteria:

* Treated at an institute where creatinine is not measured with an IDMS calibrated assay
* History of allergic reactions to computed tomography (CT) contrast, iodine or shellfish, or history of anaphylactic reaction to any food item
* Recent (last 6 months) episode of acute kidney injury, have sickle cell disease, or have current indwelling nephrostomy tubes
* Edema beyond trace edema, because this will impact iohexol equilibration and distribution
* Ascites (including pleural effusion) beyond trace ascites, because this will impact iohexol equilibration and distribution
* Whole- or part-limb amputees, because this will impact iohexol equilibration and distribution
* Inability to maintain a constant dose and schedule of anti-inflammatory agents, diuretics, angiotensin II receptor blockers (ARB) and angiotensin converting enzyme inhibitors (ACEi) for one week prior to study visit, as this impacts renal function. If the patient is on a nonsteroidal anti-inflammatory drug (NSAID), diuretic, ARB or ACEi, they are eligible as long as these agents are taken on a set schedule for 7 or more days prior to study (and not on an "as needed" basis as that can cause fluctuations in renal function)
* Inadequate venous access to obtain pharmacokinetic (PK) specimens
* Multinodular goiter, Graves' disease or autoimmune thyroiditis, per iohexol package insert (hypothyroidism is allowed)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2027-02-06 (Estimated); Study Completion 2028-02-06 (Estimated)

PRIMARY OUTCOMES:
Accuracy of achieving the targeted carboplatin area under the curve (AUC) | Up to 4 weeks
  Will be quantified by the median percentage error (PE), root-mean-squared error (RMSE), interquartile range (IQR) of the residuals, and median absolute percentage error (APE). In addition, the percentage of patients for which the observed carboplatin AUC is within 17% of target will be calculated. The actual AUC will be quantified using atomic absorption spectrophotometry.
Precision of achieving the targeted carboplatin AUC | Up to 4 weeks
  Will be quantified by the median PE, RMSE, IQR of the residuals, and median APE. In addition, the percentage of patients for which the observed carboplatin AUC is within 17% of target will be calculated. The actual AUC will be quantified using atomic absorption spectrophotometry.
Bias of the formula for estimated glomerular filtration rate (eGFR) currently in existence in patients with cancer | Up to 4 weeks
  Will be quantified by the median PE, RMSE, IQR of the residuals, and median APE will be used to assess the accuracy of each model's eGFR values for predicting measured (m)GFR. In addition, will calculate the percentage of patients for which eGFR is within 30%, 20%, and 10% of mGFR.
Precision of the formula for eGFR currently in existence in patients with cancer | Up to 4 weeks
  Will be quantified by the median PE, RMSE, IQR of the residuals, and median APE will be used to assess the accuracy of each model's eGFR values for predicting mGFR. In addition, will calculate the percentage of patients for which eGFR is within 30%, 20%, and 10% of mGFR.
Correlation between carboplatin clearance (CL) and mGFR | Up to 4 weeks
  Assessed by regression analysis. Carboplatin clearance will be derived by Empirical Bayes estimation using the POSTHOC option implemented in NONMEM. Will perform regression on the relationship between CL and mGFR. Initially this will follow a linear relationship analogous to the Calvert formula (CL = A + B* mGFR), and will test if the observed values for A and B are significantly different from those defined by Calvert as A = 25 mL/min and B = 1 (unitless). Will also perform regression by other means, e.g. after log transformation of the data, and assess if this results in a formula that performs better than the Calvert formula or the initial linear model. In addition, the impact of covariates on this relationship will be explored.

SECONDARY OUTCOMES:
Divergence of eGFR from mGFR | Up to 4 weeks
  The bias of eGFR versus mGFR will be modeled as a function of the patient's characteristics.
Success rate of achieving the target carboplatin AUC in patients in whom the carboplatin dose is capped | Up to 4 weeks
  Among patients with eGFR > 125 mL/min, precision and bias will be estimated relative to the target carboplatin AUC.
Relationship between carboplatin exposure and toxicity | Up to 4 weeks
  Will be described by the regression parameters for the estimated relationship between carboplatin AUC and platelet count, neutrophil count, and non-hematologic grade 3 toxicities.
Ability of markers in addition to creatinine in pre-treatment serum to better estimate kidney function in patients with cancer | Up to 4 weeks
  These markers will include (but are not limited to) cystatin C, beta-2-microglobulin (B2M), and beta-trace-protein (BTP). Will use these markers and patient covariates (e.g. sex, race, weight etc.) as predictors for mGFR in regression efforts.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Taylor, Principal Investigator — NRG Oncology
Locations (188):
- United States (178):
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UC San Diego Health System - Encinitas, Encinitas, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Reid Health, Richmond, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Hi-Line Sletten Cancer Center, Havre, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Clara Maass Medical Center, Belleville, New Jersey
  - Jefferson Cherry Hill Hospital, Cherry Hill, New Jersey
  - Trinitas Hospital and Comprehensive Cancer Center - Williamson Street Campus, Elizabeth, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - The Cancer Institute at Saint Francis Hospital, East Hills, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Good Samaritan University Hospital, West Islip, New York
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Vanderbilt-Ingram Cancer Center at Franklin, Franklin, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Monongalia Hospital, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Memorial Hospital of Laramie County, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Puerto Rico (10):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Puerto Rico Hematology Oncology Group, Bayamón
  - HIMA San Pablo Oncologic Hospital, Caguas
  - Doctors Cancer Center, Manatí
  - Instituto Oncologia Moderna Ponce, Ponce
  - San Juan Community Oncology Group, San Juan
  - Primary Care Physician Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan
  - San Juan City Hospital, San Juan